CLINICAL TRIAL: NCT03324932
Title: A Multicenter, Randomized, Comparative Study Regarding the Efficacy of Denosumab on Normal Bone Mineral Density in Women Receiving Adjuvant Aromatase Inhibitors for Early Breast Cancer (ENDEAVOR Trial)
Brief Title: Efficacy of Denosumab on Normal BMD in Women Receiving Adjuvant Aromatase Inhibitors for Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Principal Investigator, Hisako Ono, MD, PhD, Principal Invetstigator, Kyoto Prefectural University of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CQARD-EBS-160402; jRCTs051180211 (Registry Identifier: jRCT)
Record Dates: First submitted 2017-09-21; First posted 2017-10-30 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: bone health; hormone-sensitive breast cancer; postmenopausal; aromatase inhibitor; bone mineral density
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AI+denosumab VS only AI (Other): We compare AI intake+denosumab injection and AI intake only in patients with normal BMD to whom Letrozole or Arimidex will be administered as postoperative endocrine therapy, and we assess the efficacy of denosumab injection on bone loss by adjuvant endocrine therapy.
  Interventions: Drug: Denosumab Injection

INTERVENTIONS:
Drug: Denosumab Injection — AI intake + denosumab injection per 6 months VS only AI intake
  Other Names: pralia

SUMMARY:
This multicenter, randomized, comparative study will evaluate the efficacy of denosumab to prevent the adjuvant therapy of aromatase inhibitors-induced loss of bone mineral density (BMD) in breast cancer patients with normal BMD. Investigators will compare the inhibitory effects of denosumab on bone loss between participants with normal BMD to whom Letrozole or Arimidex will be administered as postoperative endocrine therapy for stage I-IIIA postmenopausal hormone-sensitive breast cancer and controls.

DETAILED DESCRIPTION:
Normal BMD means T score is ≥-1.0 for the lumbar vertebrae (L1-L4) and/or the femoral neck.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following items at the time of case registration:

1. Patients with infiltrative breast cancer, aged ≥20 years, meeting the following definitions:

   * Those pathologically diagnosed with stage I, II, or IIIA breast cancer (Cancer Management Regulations, 11th version)
   * Those who underwent appropriate surgery, such as mastectomy and breast-preserving surgery
2. Estrogen receptor (ER)- or progesterone receptor (PgR)-positive patients on immunohistochemical (IHC) staining
3. Females meeting one of the following criteria for menopause:

   * Those, aged ≥55 years, without menstruation
   * Those, aged <55 years, with amenorrhea for ≥12 months, or those diagnosed with menopause by attending physicians based on the FSH and estradiol levels
   * Those who underwent bilateral oophorectomy
4. Patients in whom the BMD for the lumbar vertebrae (L1-L4) on DXA before the start of this study is ≥-1.0SD of the mean value of young adult females (YAM), and the BMD for the femoral neck is ≥-1.0SD of YAM
5. Patients without lumbar vertebral or femoral fracture
6. Those with an ECOG PS of 0-2
7. Those with adequate organ functions (laboratory data within 4 weeks before case registration)

   * Leukocyte count, ≥3,000/mm3 or Neutrophil count, ≥1,500/mm3
   * AST, ALT, ≤1.5-fold of the upper limit of the institutional reference range
   * Serum creatinine, ≤1.5-fold of the upper limit of the institutional reference range
8. Case registration should be performed before the following point:Twelve weeks after the completion of surgery or postoperative chemotherapy (The completion of chemotherapy refers to the completion of the final course, involving the recovery phase.)
9. Patients with an interval of ≥4 weeks after the discontinuation of therapy with bisphosphonates (oral preparations), estrogen preparations, raloxifene, calcitonin preparations, vitamin K preparations, active vitamin D preparations, or ipriflavone preparations, which influence bones
10. Those from whom written informed consent regarding study participation was obtained

Exclusion Criteria:

Whether each patient meets any of the following items must be checked on case registration:

1. Patients in whom distant metastasis was confirmed clinically or using imaging procedures at the time of case registration
2. Those with bilateral breast cancer
3. Those for whom postoperative hormonal therapy was started before consenting to study participation
4. Those who received endocrine therapy within 52 weeks before consenting to study participation
5. Those to whom bisphosphonate preparations were intravenously administered within 52 weeks before consenting to study participation
6. Those with the following diseases that may affect DXA

   * Severe scoliosis, immobility, hyperostosis or osteosclerosis of the lumbar vertebrae, calcification of the abdominal aorta, and vertebral disease
7. Those with a history of malignant tumors other than breast cancer within 260 weeks before consenting to study participation
8. Those with dental diseases, such as infectious diseases of the teeth or jaw and tooth trauma. Those for whom tooth or jaw surgery is scheduled within 6 weeks after consenting to study participation (tooth extraction, implantation)
9. Others who are considered to be ineligible by the chief investigator

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
percentage change in the bone mineral density (BMD) for the lumbar vertebrae (L1-L4) on dual-energy X-ray absorptiometry (DXA) | 12 months after the start of this study
  The change is a value obtained by subtracting 1 from the BMD after 12 months/baseline BMD is expressed as a percentage

SECONDARY OUTCOMES:
percentage change in the BMD for the lumbar vertebrae (L1-L4) on DXA | after 2, 3, 4, and 5 years
  percentage change in the BMD for the femoral neck: After 2/3/4/5 years
percentage change in the BMD for the femoral neck | after 12 months and 2/3/4/5 years
  percentage change in the BMD for the femoral neck: After 12 months and 2/3/4/5 years
percentage change in the BMD for the radius (an ultrasonic bone densimeter is used)institutions in which ultrasonic bone densimeters are used) | after 2 and 4 weeks, every 4 weeks thereafter (for 2 years after registration)(only
  percentage change in the BMD for the radius (an ultrasonic bone densimeter is used): After 2 and 4 weeks, every 4 weeks thereafter (for 2 years after registration)(only institutions in which ultrasonic bone densimeters are used)
Changes in Ca and bone metabolism markers | after 24 weeks
  Changes in Ca (mg/dL corrected by albumin level) and bone metabolism markers such as TRAP5b, bone-specific alkaline phosphatase (BSAP), blood pentosidine) by blood sampling at every 6 months
Appearance rate of morbid fracture in all participants | up to 3 years
  Appearance rate of morbid fracture up to 3 years in all participants. Morbid fractures include all types of fractures.
Disease-free survival | at least 5 year
  Disease-free survival at the end of the study
Overall survival | at least 5 year
  Overall survival at the end of the study
Appearance of adverse events | at least 5 year
  Appearance rate of adverse events (such as hypocalcemia and necrosis of the jaw)
Quality of life (QOL) | after 24 weeks
  Quality of life(QOL), Japanese version Euro-Qol (EQ-5D-5L) evaluated by questionnaire at every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hisako Ono, PhD, Study Director — Kyoto Prefectural University of Medicine; Tetsuya Taguchi, PhD, Principal Investigator — Kyoto Prefectural University of Medicine
Locations (1):
- Hisako Ono, Kyoto, Japan

REFERENCES:
- [Background] Nakatsukasa K, Koyama H, Ouchi Y, Ono H, Sakaguchi K, Matsuda T, Kato M, Ishikawa T, Yamada K, Yoshimura M, Koizumi K, Sakurai T, Shigematsu H, Takahashi S, Taira S, Suzuki M, Narui K, Niikura N, Hasegawa Y, Miura D, Konishi E, Taguchi T; Collaborative Study Group of Scientific Research of the Japanese Breast Cancer Society. Effect of denosumab on low bone mineral density in postmenopausal Japanese women receiving adjuvant aromatase inhibitors for non-metastatic breast cancer: 24-month results. Breast Cancer. 2019 Jan;26(1):106-112. doi: 10.1007/s12282-018-0896-y. Epub 2018 Jul 27. PMID 30054855
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Sakaguchi K, Ono H, Nakatsukasa K, Ishikawa T, Hasegawa Y, Takahashi M, Niikura N, Koizumi K, Sakurai T, Shigematsu H, Takahashi S, Taira S, Suzuki M, Narui K, Miura D, Yamada K, Yoshimura M, Shioya H, Konishi E, Isao Y, Imai K, Fujikawa K, Taguchi T; Collaborative Study Group of Scientific Research of the Japanese Breast Cancer Society. Efficacy of denosumab for restoring normal bone mineral density in women receiving adjuvant aromatase inhibitors for early breast cancer. Medicine (Baltimore). 2019 Aug;98(32):e16770. doi: 10.1097/MD.0000000000016770. PMID 31393399